CLINICAL TRIAL: NCT06964269
Title: A Phase 4 Pilot Study With Extension to Assess the Use of Acthar Gel Single-Dose Pre-Filled SelfJectTM Injector in Patients With Moderate-Severe Keratitis and Autoimmune Disease and the Effect on Corneal Nerves and Neuropathic Corneal Pain
Brief Title: Use of Acthar Gel Single-Dose Pre-Filled SelfJectTM Injector in Patients With Moderate-Severe Keratitis and Autoimmune Disease
Acronym: MNK
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Toyos Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNK-MT-2024
Record Dates: First submitted 2025-04-07; First posted 2025-05-09 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Autoimmune Diseases; Dry Eye; Neurotrophic Keratitis
Keywords: Dry eye; Autoimmune; Neurotropic Keratitis
MeSH Terms: conditions — Autoimmune Diseases; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- One study arm of approximately 20 active receiving and completing active, open-label interventions. (Active Comparator): One study arm of approximately 20 active receiving and completing active, open-label interventions.
  Interventions: Drug: Acthar Gel 80 UNT/ML Injectable Solution

INTERVENTIONS:
Drug: Acthar Gel 80 UNT/ML Injectable Solution — Study intervention is twice weekly injections of Acthar Gel via single-dose pre-filled SelfJect injector for 12 weeks.

SUMMARY:
Single-site, open label pilot study of 20 autoimmune patients diagnosed with dry eye demonstrating via the proparacaine challenge some peripheral corneal pain component. At least 16 patients will receive and complete 12 weeks of 80 units of Acthar Gel to be injected subcutaneously twice weekly via Acthar Gel single-dose pre-filled SelfJectTM injector (SelfJect) to assess the effects on subjective sensation of ocular pain, conjunctival and corneal staining, in vivo assessments of corneal nerves as measured by confocal imaging, VAS scales of common neuropathic pain symptoms and comfort of SelfJect will be assessed.

DETAILED DESCRIPTION:
The primary objective of the study is to demonstrate the on-label use of Acthar Gel with SelfJect for improvement of symptoms in non-infectious keratitis related to systemic autoimmune disease and the improvement of the appearance and function of corneal nerves as visualized by confocal microscopy and demonstrated by Cochet-Bonnet) and to assess the improvement of common neuropathic corneal pain symptoms caused by dysfunctional nerves due to various autoimmune

inflammatory disease. This study will also follow patients for up to 3 years after 12 weeks of administration of Acthar Gel 80 units twice weekly to assess changes from end of treatment to end of study in visual acuity, corneal and conjunctival staining

ELIGIBILITY:
Inclusion Criteria:

1. Subject can read, understand, sign and informed consent.
2. Provision of signed and dated informed consent form and HIPPA authorization.
3. Stated willingness to comply with all study procedures and availability
4. for the duration of the study
5. Male or female aged 18-85 years.
6. Normal eyelid anatomy
7. Patients diagnosed with dry eye for at least 6 months prior to enrollment.
8. Patients with Symptom Bother score at Baseline of 50.6 or greater.
9. Patients with a diagnosis of any autoimmune disease.
10. Patients with one or more corneal neuroma as seen on baseline confocal microscopy.
11. Patients with partial or total relief of corneal pain with one drop of proparacaine over 15 minutes post-instillation.
12. No prior use of Acthar Gel SelfJect or otherwise for any indication.

Exclusion Criteria:

* 1. Have a known hypersensitivity or contraindication to the investigational product or their components.

  2. Unwilling to participate in study activities or report for study visits. 3. Current pregnancy or lactation per self-report. Patients who are unwilling to use an effective method of birth control while participating in the study and for four weeks after the last dose of study drug is administered.

  4. Use of antihistamines, mast cell stabilizers, or prescription eye drops within 24 hours prior to screening and for the study, unless the dose has been stable for 14 days.

  5. Current use of cenegermin, topical nerve growth factor or platelet rich plasma or use within the past 30 days.

  6. Treatment with another investigational drug or other intervention within 30 days of screening.

  7. Have serious or severe disease or uncontrolled medical condition that in the judgement of the investigator could confound study assessments, limit compliance, or pose safety risks.

  8. Systemic medications known to cause dry eye should not be used including antimuscarinics, antihistamines, vitamin A analogs, antianxiety agents, and others unless stable for at least 30 days.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-85
Enrollment: 20 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analog scale for injection comfort | 3 years
  To assess the severity of injection comfort in the eyes. scale ranges from 0(none) - 100(severe)
Visual Analog scale for burning | 3 years
  To assess the severity of burning in the eyes. scale ranges from 0(none) - 100(severe)
Visual Analog scale for Stinging | 3 years
  To assess the severity of stinging in the eyes. scale ranges from 0(none) - 100(severe)
Visual Analog scale for Light sensitivity | 3 years
  To assess the severity of light sensitivity in the eyes. scale ranges from 0(none) - 100(severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Toyos Clinic, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided